CLINICAL TRIAL: NCT01838135
Title: Wheelchair Self-efficacy Enhanced Training Program to Improve Wheelchair Use in Older Adults
Brief Title: WheelSeeU Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, William C. Miller, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H13-00509; H13-00509
Record Dates: First submitted 2013-03-28; First posted 2013-04-23 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Self-efficacy; Wheelchair Mobility
Keywords: wheelchair; manual wheelchair; rehabilitation; self-efficacy; older adults; feasibility; intervention; training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-based information sessions (No Intervention): Control group subjects will take part in 6 x 1.5 hour sessions of group-based information sessions facilitated by a trained instructor, consisting of topics on general wheelchair use, transportation, pain and fatigue management, nutrition, and internet resources. The instructor will be trained to not provide any training on wheelchair skills, and will be instructed to divert any wheelchair skills related questions.
- WheelSeeU Training Program (Experimental): Experimental group subjects will attend 6 x 1.5 hour training sessions (1-2 sessions/week) with a peer-Trainer. The peer-Trainer will facilitate WheelSeeU sessions and will lead participants through practice of wheelchair use goals.
  Interventions: Device: WheelSeeU Training Program

INTERVENTIONS:
Device: WheelSeeU Training Program — WheelSeeU sessions will be administered by a peer-trainer (older adult wheelchair user), who will be trained in a 2-day workshop to use social cognitive approaches (i.e. facilitating successful performance of wheelchair skills, learning through observation of peers, positive verbal reinforcement from peers and family members, and re-interpretation of physiological symptoms) to foster the improvement of self-efficacy for wheelchair use. Each WheelSeeU session will be tailored to the individual goals of participants, which will be identified during the start of each session.
  Arms: WheelSeeU Training Program

SUMMARY:
Self-efficacy predicts behavioural and rehabilitation outcomes and may be an important psychological factor for wheelchair mobility. A feasibility study will evaluate a novel self-efficacy enhanced wheelchair training intervention for older adults (WheelSeeU) to determine if: 1.WheelSeeU is feasible to administer; 2. WheelSeeU improves wheelchair use, confidence for wheelchair use, wheelchair mobility, and satisfaction with participation in older adults compared to group-based information sessions; and 3. the study design is appropriate. This feasibility study will allow for study design and protocol refinement and will provide pilot data for an experimental trial.

DETAILED DESCRIPTION:
This study will use a two-site (Vancouver and Quebec City), single blinded (Tester) RCT to compare differences in older adults' wheelchair skill with WheelSeeU versus group-based information sessions. Subjects will be randomly assigned to the experimental group (WheelSeeU) or a control group (information sessions) using a 1:1 allocation ratio between groups. To support balance between groups and blinding of assignment, a central computerized randomization process will be designed by our team statistician, with an undisclosed block size and stratified by site (Vancouver n = 20 [+4 for 20% dropout]; Quebec City n = 20 +4 ). Once subjects are enrolled, the Tester will collect baseline data and enter them into a secure database. The Site Coordinator will contact Dr. Goldsmith via telephone or email and obtain group assignment within 48 hours. Subject contact information will be forwarded to the appropriate group Trainer to arrange for an initial training session or peer support session. To address bias, subjects will be instructed not to discuss their program and the Testers (1 per site) will be blinded to group allocation. Follow-up testing will occur at immediately and 6 months post-intervention.

To mask the participants from the study objectives, participants in both the intervention and control groups will be told that the intervention is designed to improve wheelchair use. The findings from the study will be summarized and mailed to each participant upon study completion.

WheelSeeU and the control group will be held at Blusson Spinal Cord Centre, GF Strong or in the community depending on participant preference.

ELIGIBILITY:
Inclusion Criteria:

* 55 years of age or older
* live in the community
* self-propel a manual wheelchair at least 1 hour/day
* have wheelchair mobility goals
* are cognitively able to engage in the program (Modified Mini-mental Status Exam score of ≥ 24).

Exclusion Criteria:

* cannot communicate and complete study questionnaires in English
* anticipate a health condition or procedure that contraindicates training (e.g., surgery scheduled which would impair physical activity)
* have a degenerative condition that is expected to progress quickly (e.g., Amyotrophic lateral sclerosis (ALS))
* are concurrently or are planning to receive wheelchair mobility training during the period of the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Wheelchair Skills Test Version 4.1 (WST) Change | Baseline, 6 weeks, 6 month follow-up
  Wheelchair Skills Test Version 4.1 (WST) for manual wheelchair users is a standardized objective evaluation of the execution of 32 manual wheelchair skills (pass/fail) and the safety of skill execution (safe/unsafe). Total percent scores (0-100%) are calculated for both skill execution and safety. The WST was selected as the primary measure because it is a standardized tool for evaluating wheelchair capacity, the primary construct of interest.

SECONDARY OUTCOMES:
Wheelchair-use Confidence Scale (WheelCon) Version 3.0 | Baseline, 6 weeks, 6 month follow-up
  Wheelchair-use Confidence Scale (WheelCon) Version 3.0 for manual wheelchair users is a 65-item self-report scale (0-100) with documented reliability and validity. Responses indicate current level of perceived confidence (%) to navigate the physical environment in a wheelchair, perform activities in a wheelchair, problem solve, advocate for specific needs, and manage social situations and emotions. The WheelCon was selected as a secondary outcome measure because confidence for using a wheelchair has been shown to influence wheelchair skills capacity.
Wheelchair Skills Test Version 4.1 Questionnaire (WST-Q) | Baseline, 6 weeks, 6 month follow-up
  Wheelchair Skills Test Version 4.1 Questionnaire (WST-Q) for manual wheelchair users is a standardized subjective evaluation of perceived ability to execute 32 manual wheelchair skills (pass/fail). Total percent scores (0-100%) are calculated for wheelchair performance, based on whether or not the individual has successfully accomplished the skill in the past month. The WST-Q was selected as a secondary measure because it measures wheelchair skills performance, which may influence or be influenced by confidence using a wheelchair.
Life-Space Assessment (LSA) | Baseline, 6 weeks, 6 month follow-up
  Life-Space Assessment (LSA) is a 20-item questionnaire that tracks the mobility habits of wheelchair users in a continuum of environmental contexts (home; around the home; in the neighbourhood; in town; and outside of town). Participants report on their attainment of each life-space during the past 4 weeks, the frequency of attainment, and whether assistance was required. The LSA was selected as an outcome measure because it provides information about an individual's mobility habits.
Wheelchair Outcome Measure (WhOM) | Baseline, 6 weeks, 6 month follow-up
  The Wheelchair Outcome Measure (WhOM) is a client-specific measurement tool that identifies satisfaction with participation in desired activities for wheelchair users. Rates of perceived 'importance' of the goal (0-10) and 'satisfaction' with current performance of this activity (0-10) will be obtained. Scoring is calculated by multiplying 'importance' by 'satisfaction'. The WhOM was selected to obtain some information about participation goals of manual wheelchair users and to explore whether a wheelchair training intervention could influence perceived satisfaction with participation.
Late Life Function and Disability Instrument (LLFDI) | Baseline, 6 weeks, 6 month follow-up
  Late Life Function and Disability Instrument (LLFDI) is comprised of a 16-item disability component and a 40-item function component, which includes 8 items specific for individuals who use assistive devices for mobility. Participants are first asked to identify the frequency of performing life tasks using a scale ranging from 1 (never) to 5 (very often) and then asked to identify the extent that they feel limited in performing specified tasks using a scale ranging from 1 (completely) to 5 (not at all). Item responses are summed to obtain two dimension scores and four domain scores in the disability component, and one overall function score and three domain scores in the function component. The scores are then converted into interval level scores ranging from 0 to 100.
Health Utility Index Mark 3 (HUI3) | Baseline, 6 weeks, 6 month follow-up
  Health utility measurement is useful in performing cost-utility and cost-effectiveness analyses of new rehabilitation interventions. The HUI3 is a brief questionnaire that asks subjects about their health status, reflected in a single-score measure of health-related quality of life (HRQOL)

CONTACTS AND LOCATIONS:
Overall Officials: William C Miller, PhD, Principal Investigator — University of British Columbia
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Miller WC, Best KL, Eng JJ, Routhier F. Influence of Peer-led Wheelchair Training on Wheelchair Skills and Participation in Older Adults: Clinical Outcomes of a Randomized Controlled Feasibility Trial. Arch Phys Med Rehabil. 2019 Jun;100(6):1023-1031. doi: 10.1016/j.apmr.2018.10.018. Epub 2018 Nov 23. PMID 30476489
- [Derived] Best KL, Miller WC, Routhier F, Eng JJ. Feasibility of the trial procedures for a randomized controlled trial of a community-based peer-led wheelchair training program for older adults. Pilot Feasibility Stud. 2017 Jul 17;4:18. doi: 10.1186/s40814-017-0158-3. eCollection 2018. PMID 28725451
- [Derived] Best KL, Miller WC, Eng JJ, Routhier F, Goldsmith C. Randomized controlled trial protocol feasibility: The Wheelchair Self-Efficacy Enhanced for Use (WheelSeeU). Can J Occup Ther. 2014 Dec;81(5):308-19. doi: 10.1177/0008417414546743. PMID 25702375